A randomized, double-blind, placebo-controlled single and multiple dosing, escalation phase I clinical trial to investigate the safety/tolerability and pharmacokinetics of HY209 gel after transdermal administration in healthy male volunteers

Protocol No. HY209-AD (version 1.5 Date: 2019.01.20)

National Clinical Trial No. NCT03492398

Investigational Product HY209 0.05%, 0.1%, 0.3%, 0.5%

Development phase of study Phase I

Institutes Seoul National University Hospital

Sponsor Shaperon, Inc.

Protocol No.: HY209-AD Shaperon

# **■** AD Phase I Synopsis

| Study Title | A randomized, double-blind, placebo-controlled single and multiple dosing, dose escalation phase I clinical trial to investigate the safety/tolerability and pharmacokinetics of HY209 gel after transdermal administration in healthy male volunteers |
|---|---|
| Sponsor | Shaperon, Inc. |
| Institutes | Seoul National University Hospital. |
| Target disease | Atopic Dermatitis |
| Purpose | The purpose of this study is to evaluate the safety, tolerability and pharmacokinetics of HY209 gel as a possible treatment option for atopic dermatitis. |
| Study Design | Randomized, double-blind, placebo-controlled (single and multiple dosing), dose escalation phase I clinical trial |
| Study Method | Four groups (HY209 0.05%, 0.1%, 0.3%, 0.5%) of subjects, each group consisting of control 6 and placebo 2 will be randomly selected. The trial drug or placebo will be applied on the back of each subject. Subjects will be released after present tests and blood drawing. Admission Discharge Out-patient visit Out-patient visit C2) Cohort B Multiple dosing Three groups (HY209 0.05%, 0.1%, 0.3%) of subjects, each group consisting of control 6 and placebo 2 will be randomly selected. The trial drug or placebo will be applied on the back of each subject at once a day for 28 days. Subjects will visit the clinical research center to be tested |

## ■ AD Phase I Synopsis



Protocol No.: HY209-AD Shaperon

## **■** AD Phase I Synopsis

| | 2) | No okin diagona no okin domono (conve totto oto) no boin. |
|---|---|---|
| | 3) | |
| | | skin in drug-applied area which may cause the alteration of drug |
| | | absorption |
| | 4) | Those who must be capable of giving informed consent and willing |
| | | to comply with all clinic visits and study-related procedures until |
| | | study completion |
| | 1) | Those who have a history of hypersensitivity or clinically significant |
| | | hypersensitivity reactions to drugs (containing Taurodeoxycholate |
| | | component, aspirin, antibiotics, etc.) |
| | 2) | Those who have clinically significant liver, kidney, respiratory, |
| | | endocrine, neurologic diseases or hematologic diseases, mental |
| | | diseases, especially hemorrhagic diseases (hemophilia, von |
| | | Willebrand disease, etc.), cardiovascular diseases (coronary artery |
| | | diseases, congestive heart failure, arrhythmia, cerebrovascular |
| | | diseases, etc.) or who have a history of those diseases |
| | 3) | Those who have clinical symptoms suspected of acute infectious |
| | 3) | · |
| | | disease within 2 weeks before the schedule date of the first |
| | | administration, or whose temperature measured by the screening |
| | | test was 38°C or higher |
| Exclusion | 4) | Those who have taken any ETC medicines, herbal medicines, crude |
| Criteria | | drugs within 2 weeks before the scheduled date of administration of |
| | | medicines for clinical trials, or OTC medicines or vitamin |
| | | preparations within 1 week (if all other selection / exclusion criteria |
| | | are met. The researcher should consult with the sponsor to |
| | | determine whether it is appropriate to take the subject into the trials, |
| | | considering the safety of the subject or the effect on overall clinical |
| | | trial results.) |
| | 5) | Those who have a history of substance abuse, or positive urine |
| | , | screening tests (cannabinoid, opiates, amphetamine, cocaine, |
| | | barbiturate, benzodiazepine) |
| | 6) | Those who have a history of smoking within 3 months (However, if |
| | 5, | they quit smoking three months before the first scheduled |
| | <b>7</b> \ | medication, they are eligible for selection) |
| | 7) | Those who have been found to be positive in serological tests (HBs |

Protocol No.: HY209-AD Shaperon

### AD Phase I Synopsis

antigen, HCV antibody and HIV antibody) 8) Those who drink continuously (above 21 units / week, 1 unit = 10 g of pure alcohol) 9) Those who have been taking medicines by participating in other clinical trials or bioequivalence studies within 3 months prior to the date of first dosing (the time from the date of the previous clinical trial will be based on the date of administration of each relevant clinical trial drug, If the half-life of a test drug taken in a clinical trial is more than two weeks, it may be attained more than five times the expected half-life of the test drug.) 10) Those who have been bleeding, blood drawings or blood donation of 400mL or more within 8 weeks before the scheduled date of administration of the drug for clinical trials 11) Those who have vital signs measured at sitting postion after the break for more than 3 minutes, Low blood pressure (systolic blood pressure < 90 mmHg, diastolic blood pressure < 50 mmHg) High blood pressure (systolic blood pressure greater than 150 mmHg, diastolic blood pressure greater than 100 mmHg) 12) Test subjects who are deemed unsuitable for participating in clinical trials due to clinical laboratory tests, ECG results, or other reasons **Primary Outcome Measures** 1) Safety and tolerability assessment Adverse events, physical symptoms, vital signs, physical test, **Outcome** electrocardiography, clinical laboratory test, local stimulation Measures assessment, numerical plan rating scale **Secondary Outcome Measures** Pharmacokinetics Cmax, ss, Cmin, ss, AUCinf, T, ss, Tmax, ss, t<sub>1/2</sub>, ss, CL/F

#### CONFIDENTIAL